CLINICAL TRIAL: NCT01236924
Title: Effectiveness of Global Postural Reeducation in Patients With Chronic Symptomatic Lumbar Disc Herniation
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Universidade Gama Filho (Other)
Purpose: Treatment
Other Study IDs: 112.2010
Record Dates: First submitted 2010-11-08; First posted 2010-11-09 (Estimated); Last update posted 2010-11-09 (Estimated); Status verified 2010-11

CONDITIONS: Lumbar Disc Herniation.
MeSH Terms: conditions — Intervertebral Disc Displacement

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Lifestyle counseling (Experimental)
  Interventions: Other: Global postural reeducation

INTERVENTIONS:
Other: Global postural reeducation

SUMMARY:
Slipped disc is the rupture of the fibrous ring, with subsequent displacement of the nucleus pulposus in intervertebral spaces, which may cause compression of nerve structures. It is estimated that 2-3% of the population have taken with this process, whose prevalence is 4.8% in men and 2.5% in women over 35 years. Thus, the purpose of this study is to verify the effectiveness of global postural reeducation in patients diagnosed with chronic symptomatic lumbar disc herniation with the application of a randomized controlled trial. Will be measured pain, disability and functional flexibility.

ELIGIBILITY:
Inclusion Criteria:

Patients diagnosed with chronic symptomatic lumbar disc herniation

Exclusion Criteria:

Patients who work with severe overloading of the spine, patients with central neurological pathology, wheelchair users, patients who use bracing and support those who submit two consecutive absences to the treatment

Ages: 25 Years to 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Dates: Start 2011-01

CONTACTS AND LOCATIONS:
Locations (1):
- Gama Filho University, Rio de Janeiro, Rio de Janeiro, Brazil